CLINICAL TRIAL: NCT05352568
Title: Is Cognitive Training an Option? Understanding the Feasibility of Cognitive Training With Individuals Living With Schizophrenia
Brief Title: Is Cognitive Training an Option?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliant International University (Other)
Responsible Party: Principal Investigator, Andre Pierre Longino, M.A., Researcher, Alliant International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2105211050
Record Dates: First submitted 2021-06-14; First posted 2022-04-29 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Schizophrenia; Schizoaffective; Cognition
Keywords: Schizophrenia; Schizoaffective; Cognition; Social Cognition; Psychosocial Function
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Pre-test/post-test pre-experimental design with convenience and snowball sampling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Group (Experimental): Computer Cognitive-Based Training
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Cognitive Training — Computer-Based Cognitive Training from BrainHQ (Posit Science)

SUMMARY:
The purpose of the study is to evaluate the feasibility of implementing cognitive training with 40 patients living with schizophrenia and schizoaffective disorder. The study aims to explore if cognitive training as an intervention can improve cognition, symptomology, social cognition, and psychosocial function which has been determined through literature to be impacted within this population. The results of this study will help shed light on utilizing additional resources to aid in decreasing relapse and continued hospitalizations.

DETAILED DESCRIPTION:
After being selected for this study based on a screening survey, participants will be asked to fill out a demographic questionnaire, the Multidimensional Schizotypy Scale - Brief Version (MSS-B), the Montreal Cognitive Assessment (MoCA), the Davos Assessment of Cognitive Biases Scale (DACOBS), and the Illness Management and Recovery Scale - Consumer Self-Rating, IMRS. The measurements evaluate different aspects of severe mental illness which are often challenges. This will take approximately: the screener questionnaire (2-3 minutes), demographic questionnaire (3-5 minutes), MSS-B (38 questions: 10-15 minutes), MoCA (10-15 minutes), DACOBS (42 questions: 15-20 minutes), and IMS (15 questions: 5 to 15 minutes)- Total Maximum Time is 63 minutes. After all, measurements are completed, the participants will be introduced to the BrainHQ program the following week. The participants will begin the selected cognitive training module 3 times a week (Mon, Wed, and Fri), 60 minutes per session for a total of 180 minutes per week. The participants will have a total of 24 sessions over the course of 8 weeks, for a total of 1,440 minutes of cognitive training over the course of this feasibility study. A process questionnaire on the acceptability/ feasibility of the cognitive training program will be administered after the first session, then the middle progress point (4th week), and at the end of the program (8th week) (2-3 minutes). Upon completion of the cognitive training, the participants will retake each measurement (MSS-B, MoCA, DACOBS, and IMRS)-Total Maximum Time is 55 minutes. There is minimal to no risk in this study. Participants will continue their prescribed treatment plan with the addition of the cognitive training which is computerized and takes the form of simulated games with an attended purpose. Participants will continue to be monitored by their providers and staff will continue to evaluate participants for changes in baseline behavior on a daily basis during the course of the study. The plan analysis for this study will be a MANOVA and Correlations. Confidentiality of research records and data will be protected in accordance with the Alliant International University Institutional Review Boards policies, and procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* A diagnosis of schizophrenia or schizoaffective disorder
* All genders
* All sexual orientations
* All class/ social-economic status
* All ethnicities

Exclusion Criteria:

* An inability to understand the consent process and/or provide assent
* Inability to understand the assent form/process
* Not being a fluent English speaker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 10-15 minutes
  A quick screening tool for mild cognitive impairments (MCI) and early Alzheimer's dementia.

SECONDARY OUTCOMES:
Davos Assessment of Cognitive Biases Scale (DACOBS) | 15-20 minutes
  A self-report measure of cognitive biases and cognitive limitations that contributes to psychosis.
Illness Management and Recovery Scale - Consumer Self-Rating, IMRS | 5-15 minutes
  A psychosocial functioning assessment for individuals with schizophrenia.
Multidimensional Schizotypy Scale - Brief Version (MSS-B) | 10-15 minutes
  A symptomology assessment with a subscale consisting of positive, negative, and disorganized dimensions of schizotypy.

CONTACTS AND LOCATIONS:
Locations (1):
- View Heights Convalescent Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No